CLINICAL TRIAL: NCT04858568
Title: PROSECO - A UK Multicentre Prospective Observational Study Evaluating COVID-19 Vaccine Immune Responses in Lymphoid Cancer
Brief Title: Immune Responses to COVID-19 Vaccination in Lymphoma Patients
Acronym: PROSECO
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CAN1612
Record Dates: First submitted 2021-04-22; First posted 2021-04-26 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Classical Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Primary Mediastinal B Cell Lymphoma; High-grade B-cell Lymphoma; Burkitt Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Lymphoplasmacytic Lymphoma; Nodular Lymphocyte Predominant Hodgkin Lymphoma; Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Burkitt Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma Serum Peripheral blood mononuclear cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hodgkin lymphoma: Diagnoses:
  Hodgkin lymphoma (classical Hodgkin lymphoma)
- Aggressive B-NHL: Diagnoses:
  Aggressive B-NHL (E.g. Diffuse large B-cell lymphoma, primary mediastinal B-cell lymphoma, high-grade B-cell lymphoma, Burkitt lymphoma, de novo transformed lymphoma, follicular lymphoma grade 3b)
- Indolent B-NHL: Diagnoses:
  Indolent B-NHL (E.g.follicular lymphoma grades 1-3a, mantle cell lymphoma, marginal zone lymphoma, chronic lymphocytic leukaemia/small lymphocytic lymphoma, lymphoplasmacytic lymphoma, nodular lymphocyte predominant Hodgkin lymphoma)
- Peripheral T/NK-cell: Diagnoses:
  Peripheral T/NK-cell lymphomas (any mature T/NK cell malignancy)

SUMMARY:
This prospective observational study aims to evaluate the robustness and persistence of immune responses to vaccination, define factors associated with impaired immune responses and assess the incidence of COVID-19 infections in vaccinated individuals. To do this, we will collect peripheral blood from patients with lymphoid cancers before and after their COVID-19 vaccination. The blood will be explored in the laboratory for antibodies to SARS-CoV-2 and T-cell responses to the spike protein. Detailed clinical information will also be collated on about their cancer and treatment.

ELIGIBILITY:
INCLUSION CRITERIA

1. Patients having a confirmed diagnosis of either:

   A) Hodgkin lymphoma B) Aggressive B-cell lymphoma (e.g. Burkitt's lymphoma, diffuse large B-cell lymphoma, grade 3b follicular lymphoma, de novo transformed follicular lymphoma) C) Indolent B-cell lymphoma (e.g. all grades of follicular lymphoma except grade 3b, marginal zone lymphoma, lymphoplasmacytic lymphoma, chronic or small lymphocytic lymphoma, mantle cell lymphoma) D) Mature T/NK-cell malignancy (any subtype)
2. Patient must be ≥ 18 years.
3. Patients will have provided written Informed Consent.

EXCLUSION CRITERIA

1) Serious medical or psychiatric illness likely to affect participation or that may compromise the ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a confirmed lymphoma diagnosis who is under the care of a secondary or tertiary referral centre.
Sampling Method: Non-Probability Sample
Enrollment: 592 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Serum IgG levels against SARS-CoV-2 post-COVID-19 vaccination and change over time. | 12 months
  To evaluate the robustness and persistence of anti-S IgG levels.

SECONDARY OUTCOMES:
Comparison between SARS-CoV-2 IgG responses with clinical parameters. | 12 months
  Correlation between anti-S IgG between different lymphoma subtypes and the impact of treatment.
Symptomatic COVID-19 with positive SARS-CoV-2 PCR results. | 12 months
  To assess the incidence of symptomatic, virologically proven COVID-19 in vaccinated individuals within 12 months of vaccine administration.

CONTACTS AND LOCATIONS:
Locations (9):
- United Kingdom (9):
  - Bedfordshire Hospitals NHS Foundation Trust, Bedford, Bedfordshire
  - Portsmouth Hospitals University NHS Trust, Portsmouth, Hampshire
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Wye Valley NHS Trust, Hereford, Herefordshire
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich, Norfolk
  - Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear

REFERENCES:
- [Derived] Lim SH, Stuart B, Joseph-Pietras D, Johnson M, Campbell N, Kelly A, Jeffrey D, Turaj AH, Rolfvondenbaumen K, Galloway C, Wynn T, Coleman AR, Ward B, Long K, Coleman H, Mundy C, Bates AT, Ayres D, Lown R, Falconer J, Brake O, Batchelor J, Willimott V, Bowzyk Al-Naeeb A, Robinson L, O'Callaghan A, Collins GP, Menne T, Faust SN, Fox CP, Ahearne M, Johnson PWM, Davies AJ, Goldblatt D. Immune responses against SARS-CoV-2 variants after two and three doses of vaccine in B-cell malignancies: UK PROSECO study. Nat Cancer. 2022 May;3(5):552-564. doi: 10.1038/s43018-022-00364-3. Epub 2022 Mar 24. PMID 35332334